CLINICAL TRIAL: NCT03066336
Title: A Pilot Evaluation of the Effect of the Erchonia LunulaLaser for the Treatment of Toenail Onychomycosis
Brief Title: A Study to See if Low Level Laser Light Can Help to Treat Toenail Fungus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting subjects
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC_LL_MYC_PS
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Onychomycosis of Toenail

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Erchonia LunulaLaser (Experimental): The Erchonia LunulaLaser emits both red light (635 nm) and blue light (405 nm) to the affected toenail for 12 minutes per treatment for 4 treatments, each treatment one week apart.
  Interventions: Device: Erchonia LunulaLaser

INTERVENTIONS:
Device: Erchonia LunulaLaser — Active Low Level Laser Light Therapy

SUMMARY:
The purpose of this study is to determine whether low level laser therapy (LLLT) using the Erchonia LunulaLaser device is effective in clearing toenails with onychomycosis.

DETAILED DESCRIPTION:
Nail onychomycosis, or fungus infection, is typically caused by a fungus called dermatophytes, but may also be caused by yeasts and molds. These microscopic organisms invade the skin through tiny invisible cuts or through a small separation between the nail and the nail bed. Under conditions of warmth and moisture, the fungi grow and spread. The infection begins as a white or yellow spot under the tip of the nail, and as it spreads deeper into the nail, causes unsightly and potentially painful nail discoloration, thickening and the development of crumbling edges. Onychomycosis occurs more commonly in toenails than in fingernails because toenails are often confined in a dark, warm, moist environment inside shoes where fungi can thrive. Toenail fungus affects approximately 23 million people in the US - about 10% of all adults.

Potential complications of onychomycosis include pain in the nails, permanent damage to the nails, development of other serious infections that can spread beyond the feet for individuals with a suppressed immune system due to medication, diabetes or other conditions, such as leukemia and AIDS.

Nail fungus can be difficult to treat, and repeated infections are common. Currently available treatments for onychomycosis include oral antifungal medications, antifungal lacquer, and topical medications, surgical nail removal and photodynamic therapy. There is no perfect cure for toenail fungus. Even the most effective oral medications are successful only about half of the time, and topical medications are successful less than 10% of the time. Recently, research has found laser therapy to show promise as a novel alternative treatment for toenail onychomycosis. Unlike medication-driven treatments for toenail fungus which can have many side effects including serious ones such as liver toxicity, laser therapy presents minimal to no risk of side effects. Laser therapy is applied to toenail onychomycosis by shining a laser light through the toenail into the tissue below. The laser light vaporizes the fungus while leaving the skin and surrounding healthy tissue unharmed.

Low level laser therapy operates under the principle of photochemistry with a photoacceptor molecule absorbing the emitted photons and inducing a biological cascade. Like our eukaryotic cell, fungi contain the highly complex organelle the mitochondria, which is responsible for the manufacturing of the energy molecule adenosine triphosphate (ATP). Within the inner mitochondrial membrane is cytochrome c oxidase, an identified photoacceptor molecule. It is believed that laser therapy could perhaps provide a means to photo-destroy the fungi responsible for onychomycosis (OM) by inducing the release of highly reactive superoxides. Moreover, laser therapy has been shown to promote superoxide dismutase (SOD), a process responsible for the destruction of foreign invaders. Extracellular release of low levels of mediators associated with SOD can increase the expression of chemokines, cytokines, and endothelial leukocyte adhesion molecules, amplifying the cascade that elicits the inflammatory response. The physiologic function of hydrogen peroxide, superoxide anion, and hydroxyl free radical is to destroy phagocytosed microbes. By enhancing the natural processes of the immune system and impacting the structural integrity of the fungi strain, it is believed that laser therapy may provide a means for clinicians to effectively treat OM without the onset of any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Visual clinical presentation of onychomycosis in the target great toenail is distal subungual onychomycosis (DSO), visualized as a nail with normal surface texture and thickness but variable "bays" of white nail that extend from the distal nail tip proximally into the area of the nail bed
* Clinical involvement of onychomycosis in the target toenail is up to 60%
* Confirmation of the presence of fungal infection through a positive KOH stain finding and a positive fungal culture finding
* Identification through fungal culture of the growth of Trichophyton rubrum (T. rubrum) or other common dermatophyte or C. albicans or mixed dermatophyte/Candida infection. In the event of the KOH stain and the fungal culture provide conflicting results, i.e., one is positive and the other negative, resolution may be obtained by a second negative fungal culture finding from a nail clipping from the same nail
* Subject is willing and able to refrain from employing other (non-study) treatments (traditional or alternative) for his or her toenail onychomycosis throughout study participation.
* Subject is willing and able to refrain from the use of nail cosmetics such as clear and/or colored nail lacquers throughout study participation

Exclusion Criteria:

* Visual clinical presentations of onychomycosis in the target great toenail that are inconsistent with the clinical presentation of distal subungual onychomycosis (DSO), in whole or in part (i.e. indicative of mixed etiology); specifically proximal subungual onychomycosis (PSO); superficial white onychomycosis (SWO); complete dystrophy; other nail changes.
* Identification through fungal culture of the growth of a rare fungal species (i.e. not Trichophyton rubrum (T. rubrum) or other common dermatophyte or C. albicans or mixed dermatophyte/Candida infection) or non-fungal organisms such as mold or bacteria
* Less than 2mm clear (unaffected) nail plate length beyond the proximal fold
* Presence of dermatophytoma (thick masses of fungal hyphae and necrotic keratin between the nail plate and nail bed)
* Infection involving lunula e.g., genetic nail disorders, primentary disorders
* Severe plantar (moccasin) tinea pedis
* Psoriasis of the skin and/or nails, lichen planus, or other medical conditions known to induce nail changes
* Onychogryphosis
* Trauma from ill-fitting shoes, running, or overly-aggressive nail care
* Previous toenail surgery
* Uncontrolled diabetes mellitus
* Peripheral vascular disease
* Recurrent cellulitis
* Lymphatic insufficiency
* Immune compromise (whether due to underlying medical disorders or immuno-suppressive treatments)
* Other compromised states of health
* Known photosensitivity disorder
* Use of oral antifungal drugs in the prior 6 months
* Use of topical treatment of the skin or nails within the prior 2 months
* Any abnormality of the toenail that could prevent a normal appearing nail from occurring if clearing of infection is achieved.
* Current trauma, open wound on or about the treatment area
* Deformity of the target toe/toenail secondary to fungal infection/onychomycosis due to prior injury, surgical procedures or another medical condition
* Pregnant or planning pregnancy prior to the end of study participation
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to follow study subject requirements and/or record the necessary study measurements
* Involvement in litigation and/or receiving disability benefits related in any way to the parameters of the study
* Participation in a clinical study or other type of research in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Percent (%) of toenails attaining mycologic cure at study endpoint | 3 months
  Mycologic cure is defined as both negative Potassium Hydroxide (KOH) and negative Fungal Culture results, or two serial negative Fungal Culture results.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Tosti, MD, Principal Investigator; Ted Rosen, MD, Principal Investigator — unaffilliated
Locations (1):
- University Of Miami Department of Dermatology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No